CLINICAL TRIAL: NCT03556462
Title: Increasing Sleep Health Literacy: A Social Ecological Approach
Brief Title: Sleep Health Literacy in Head Start
Acronym: SLEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Karen Bonuck, Professor, Albert Einstein College of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2014-3031; R01HD082129 (NIH)
Record Dates: First submitted 2018-05-18; First posted 2018-06-14 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Sleep

STUDY DESIGN:
Intervention Model Description: Stepped wedge cluster RCT Participating agencies (n=7) were randomly assigned to 'wedge 1' or 'wedge 2': Wedge 1 agencies will begin the intervention in Fall 2018 and Wedge 2 agencies will begin the intervention in Spring 2019.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Health Interventions (Experimental): Sleep Health Interventions:
  Parents- a) invited to 1 hour workshop about healthy sleep, b) invited to attend a brief (app. 20 minute) Sleep Health Flipchart education either 1-on-1 or in a small group.
  Children: exposed to 2 week 40min/day healthy sleep curriculum in the classroom.Agency: Video and print material
  Interventions: Other: Sleep Health Education
- Control Period (No Intervention): No Intervention, but data collection

INTERVENTIONS:
Other: Sleep Health Education — Parents and children receive sleep health education
  Arms: Sleep Health Interventions

SUMMARY:
Conduct Sleep Health Literacy RCT- Using a stepped wedge randomized design, investigators will enroll 540 parent-child dyads from 7 Head Start agencies in New York. Agencies cross-over from control to intervention. Outcomes are a) child sleep duration, b) parent knowledge, attitudes, self-efficacy and behavior, c) child sleep difficulty and d) classroom climate. Invesetigators will compare intervention vs. control data across agencies and pre/post data within agency, with parental health literacy as a moderator. Investigators will collect process and fidelity data.

DETAILED DESCRIPTION:
Abstract: Inadequate and/or poor quality sleep in early childhood impairs social-emotional and cognitive function (via effects on the developing brain), and markedly increases obesity risk (via hormonal and endocrine effects). Short sleep duration, behavioral sleep problems and sleep-disordered breathing peak at 20%-50%, during the preschool years (ages 3-5). Healthy sleep habits increase sleep duration and prevent behavioral sleep problems. Awareness of sleep-disordered breathing symptoms leads to timely treatment for it. Despite ample data on sleep problems "…much less work has been done on effective strategies to promote sleep as a healthy behavior (CDC 2013)". This study's overarching goal is to empower families of preschool children with the knowledge and skills needed for healthy sleep, and to recognize a sleep problem. It builds on work in Head Start, an early childhood education (ECE) program for disadvantaged preschool children and their families: The team's Early Childhood Sleep Education Program (ECSEP™) educates Head Start teachers, children, and parents about healthy sleep in a way they can process and understand. In a randomized controlled trial, the children in the ECSEP group slept 30 minutes longer/night. As well, our UCLA Health Care Institute's structured approach to low literacy health training in Head Start (to reduce ER visits, obesity, etc.) has reached >100,000 families. The proposed study will implement a Social-Ecological web of multi-level interventions to reinforce the ECSEP, and to promote healthy sleep throughout ECE. Within Head Start, the team will create new delivery platforms (print & video, family visits) that 'amplify' the ECSEP. Beyond Head Start, the team will educate communities, and partner with stakeholders on strategies designed to embed 'sleep health literacy' in ECE policy. This project will: 1) Adapt sleep education material into additional multi-media formats, and; apply the Health Care Institute model to train Head Start staff to mount interventions and collect data. 2) Enroll 540 parent-child dyads from 7 Head Start agencies in New York in a stepped wedge randomized controlled trial. Investigators will analyze trial effects on primary outcomes: a) child sleep duration, b) parent knowledge, attitudes, self-efficacy and behavior, and c) child sleep difficulties. 3) Assess the feasibility of screening and guidance for sleep problems (vs. sleep health) for a future efficacy study. Secondary outcomes are: classroom behaviors, policy change, and process data. Poor sleep in early development has ramifications for years to come, perhaps through adulthood. Head Start serves low-income, mainly racial-ethnic minority families, in whom sleep health disparities are greatest-- but are modifiable. This study joins together proven methods of delivering health literacy (Health Care Institute) and sleep health (ECSEP) programs in Head Start. Intervening at every level of the Social-Ecological model maximizes the study's reach and sustainability. Integrating sleep health literacy into ECE nationwide could ultimately benefit upwards of 4 million children. The potential impact upon human health is far-reaching.

ELIGIBILITY:
Inclusion Criteria:

1. Attends 3-year old Head Start class at site for 2018-2019 school year
2. English or Spanish
3. Family affirms that plans are for child to remain at site for duration of school year (per screener item)
4. Respondent affirms that they are regularly involved in the child's bedtime routine (per screener item)

Exclusion Criteria:

* Child not age-eligible (see above)
* Family not language eligible (see above)
* Family not planning to remain for duration of 2018-19 school year

Ages: 3 Years to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 538 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2022-02-03 (Actual)

PRIMARY OUTCOMES:
Child Sleep Duration: Intervention vs. Control (Total) | 9 months
  The primary outcome is differences between Intervention vs. Control periods (per stepped wedge design) weeknight sleep: Sunday-Thursday bedtimes and Monday-Friday wake-times. Agency staff will distribute and collect sleep logs from parent participants at 5 points: 1 week pre/post the 2 "cross-overs" and at final follow-up. Analyses will be based upon weeknight (Sun-Thurs) sleep duration from sleep logs, assessed in minutes.
  Hypothesis: longer sleep duration for Intervention vs. Control periods

SECONDARY OUTCOMES:
Child Sleep Duration: >30 Minutes | 9 months
  Hypothesis: Intervention group will sleep >= 30 minutes longer than Controls difference in duration between Intervention vs. Control periods
Child sleep difficulties | 12 months
  Tayside Children's Sleep Questionnaire- This simple 10-item tool detects 'settling' difficulties (e.g., getting to/staying asleep) in 1-5 year olds. Nine items, scored on a 5-point scale, refer to the past 3 months: a score of > 8/36 indicates a mild/moderate settling difficulty. The last (yes/no) item asks if the child has a sleep problem. hypothesize: a) lower mean Tayside scores for Intervention vs. Control periods, b) a lesser likelihood of Intervention vs. Control scores above the criterion indicative of mild/moderate difficulties (> 8/36) and c) lower rates of parents reporting a sleep problem (Yes/No) in Intervention vs. Control periods.
Parent KASB (Knowledge/Attitudes/Self-Efficacy/Beliefs) | 12 months
  Parents rate agreement with items on a 5-point scale. Knowledge items (n=12); Attitude items (n=5); Self-efficacy items (n=7) and Belief items (n=2) query the value of a regular bedtime and bedtime routine. There is one multiple-choice item about how much sleep a preschooler needs.
  Hypotheses: a) higher KASB total scores for Intervention vs. Control phases, and b) higher scores for each of the Knowledge, Attitudes, Self-Efficacy, and Behavior domains for Intervention vs. Control phases. As descriptive data, repeat analyses will be conducted for pre/post the ECSEP within each agency.
Child Sleep Duration: 1 Year Follow-Up | 12 months
  Hypothesis: Intervention group will sleep >= 15 minutes longer than Controls at 1 Year Follow-Up
Classroom Climate | 9 months
  Investigators will collect a measure of classroom climate, reflecting teacher-child interactions:
  ● Classroom Climate- the Classroom Assessment Scoring System (CLASSTM) is an evidence-based tool developed by the NIH. Data are collected quarterly by certified observers. We will analyze CLASS data for: Positive Climate, Negative Climate, and Behavior Management. Scores range from 1-7: Low (1-2), Medium (3-4) and High (5-7).
  It is hypothesized that CLASS scores (or their equivalent) for Positive Climate, Negative Climate, and Behavior Management will differ significantly for Intervention vs. Control periods at the classroom, site, and agency levels.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Bonuck, PhD, Principal Investigator — Albert Einstein College of Medicine
Locations (7):
- United States (7):
  - Yeled v"Yalda Early Childhood Center, Inc., Brooklyn, New York
  - Committee for Early Childhood Development D.D.C. incl, Hollis, New York
  - East Harlem Council for Human Services, Inc., Manhattan, New York
  - Cattaraugus and Wyoming Counties Project Head Start, Olean, New York
  - Agri-Business Child Development, Schenectady, New York
  - Kingsbridge Heights Community Center, The Bronx, New York
  - Family Services of Westchester, White Plains, New York

REFERENCES:
- [Derived] Bonuck K, Collins-Anderson A, Schechter CB, Felt BT, Chervin RD. Effects of a Sleep Health Education Program for Children and Parents on Child Sleep Duration and Difficulties: A Stepped-Wedge Cluster Randomized Clinical Trial. JAMA Netw Open. 2022 Jul 1;5(7):e2223692. doi: 10.1001/jamanetworkopen.2022.23692. PMID 35881396
- [Derived] Bonuck K, Collins-Anderson A, Ashkinaze J, Karasz A, Schwartz A. Environmental Scan of Sleep Health in Early Childhood Programs. Behav Sleep Med. 2020 Sep-Oct;18(5):598-610. doi: 10.1080/15402002.2019.1640222. Epub 2019 Jul 18. PMID 31318273